CLINICAL TRIAL: NCT06425822
Title: Characterization of Left Atrial Substrate in Patients With Ventricular Arrhythmias
Acronym: CLASS-VA
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Andrea Sarkozy, Clinical Professor, Universitair Ziekenhuis Brussel
Other Study IDs: EC-2023-281
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Atrial Remodeling
MeSH Terms: conditions — Atrial Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left atrial mapping group in patients without atrial fibrillation: Inclusion criteria:
  * Age ≥ 18 years old.
  * Absence of a prior history of atrial fibrillation or flutter.
  * Patients presenting for ablation of any ventricular tachycardia related to structural heart disease or any ventricular arrhythmia with a CHA2DS2-VASc score ≥ 2.
  Exclusion criteria:
  * Presence of thrombus in the left atrial appendage.
  * Complications related to the index procedure.
  * Insufficient quality of the left atrial electroanatomical map.
  Interventions: Diagnostic Test: Left atrial electroanatomical mapping

INTERVENTIONS:
Diagnostic Test: Left atrial electroanatomical mapping — Left atrial electroanatomical mapping (substrate and functional mapping)

SUMMARY:
The goal of this observational study is to analyze the characteristics of left atrial electroanatomical maps in patients without a history of atrial fibrillation but with a high clinical risk of developing it, as indicated by the presence of structural heart disease or a CHA2DS2-VASc score ≥ 2 points. The study cohort will be compared to a historical cohort of patients with diagnosed atrial fibrillation in a propensity-matched fashion.

The main questions it aims to answer are:

* Are the left atrial electroanatomical changes a consequence or a precursor to the development of atrial fibrillation?
* Are the left atrial electroanatomical findings different between patients with atrial fibrillation and those at high risk of developing it?
* What is the prognostic impact of left atrial pathologic changes in patients without diagnosed atrial fibrillation in terms of cardiovascular outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Absence of a prior history of atrial fibrillation or flutter.
* Patients presenting for ablation of any ventricular tachycardia related to structural heart disease or any ventricular arrhythmia with a CHA2DS2-VASc score ≥ 2.

Exclusion criteria:

* Presence of thrombus in the left atrial appendage.
* Complications related to the index procedure.
* Insufficient quality of the left atrial electroanatomical map.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing ventricular arrhythmias ablations in whom transeptal access is needed for the ablation of the targeted arrhythmia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Substrate characterization of the left atrium. | 18 months
  Substrate characterization will involve measuring Low Voltage (LV) and Transition Voltage (TV) Zones (LV zone voltage cut-off of <0.5mV; TV zone voltage limits within 0.5 and 1mV). These zones will be considered if they encompass an area of at least 1cm², containing ≥3 neighboring points within ≤10mm distance. The total LVZ and TVZ surfaces will be expressed as a percentage relative to the total surface area of the left atrium (excluding the pulmonary veins and the mitral annulus).
  A comparative analysis of substrate characteristics will be conducted between two groups: the study group (comprising patients without atrial fibrillation but at risk of developing it) and the control group (a historical cohort of patients with known atrial fibrillation).
Functional characterization of the left atrium. | 18 months
  Functional analysis will rely on identifying deceleration zones characterized by isochronal crowding, defined as having ≥3 isochrones within a 1cm radius, using an 8-color scale of left atrial isochronal activation mapping.
  A comparative analysis of functional characteristics will be conducted between two groups: the study group (comprising patients without atrial fibrillation but at risk of developing it) and the control group (a historical cohort of patients with known atrial fibrillation).

OTHER OUTCOMES:
Incidence of atrial fibrillation during follow-up. | 12 months
  Episodes diagnosed via a single-lead ECG tracing or a complete 12-lead ECG lasting at least 30 seconds, or AHRE episodes detected by any cardiac implantable electronic device (CIED), lasting at least 5 minutes.
Incidence of myocardial infarction during follow-up | 12 months
  Only type 1 myocardial infarctions, those related to acute coronary obstruction, will be considered.
Incidence of stroke during follow-up | 12 months
  Stroke will be defined as any objective evidence of permanent brain, spinal cord, or retinal cell death resulting from a vascular cause, substantiated by pathological or imaging evidence, with or without accompanying clinical symptoms.
Incidence of transient ischemic attack incidence during follow-up | 12 months
  Transient ischemic attack will be defined as a sudden, focal neurological deficit of presumed vascular origin lasting less than 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sarkozy, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided